CLINICAL TRIAL: NCT04330352
Title: "STOP Touching Your Face": a Randomized Controlled Trial of Brief Mindfulness-based Intervention
Brief Title: Mindfulness-based "STOP (Stop, Take a Breath, Observe, Proceed) Touching Your Face" Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Psychiatrist, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020S001
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Face-touching Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based "STOP touching your face" intervention (Experimental): Eligibility participants who are allocated to the intervention group will be required to find a time to monitor and record their behavior of hand-to-face contacts, including the frequency and length (in second) of face-touching in any of the mucosal area (eyes, nose, mouth) and nonmucosal area (ears, cheeks, chin, neck, forehead, hair) during a 60-minute period. Then, they will receive the online mindfulness-based "STOP touching your face" program. Each participant will be required to practice this technique until they feel confident and natural. The systematic review showed the efficacy of single session of brief MBIs, the average length was 15 minutes, ranged from less than 5 to 25 min. Thus, the requirement practice time will be at least 15 minutes (excluding the time of reading the text and the first time of listening to the audio). Later (at least 1-hour interval), they will be asked to self-monitor and report their one-hour face-touching behavior again.
  Interventions: Behavioral: Mindfulness-based "STOP touching your face" practice
- Contron information intervention (No Intervention): Participants who allocate to the control group will only receive information to thank them and encourage them to complete the study. They will receive "STOP touching your face" program after the end of this study. The repeat measurement of the face-touching behavior will be in at least 1-hour interval.

INTERVENTIONS:
Behavioral: Mindfulness-based "STOP touching your face" practice — 1. Remind yourself to STOP. Whatever you are doing in this moment (e.g. touching your month, pinching your nose, rubbing your eyes, resting your chin on your hands), pause for a minute. 2. Take a deep breath. This reconnects you with your body. Pay attention to your breathing and just allow yourself to continue to breathe normally and naturally. 3. Observe what is happening for you in this moment-including thoughts, feelings, and emotions (e.g. feel distracted, anxious or nervous?). What do you notice in your body (e.g. feel itchy or tingling on any part of your face)? You can be aware of anything: posture, sensations, tension in your body, or, once again, your breath. You might notice the sound around you. You might even notice your thoughts or emotions. 4. Proceed with whatever you were doing before you came to a STOP or something that you want to do in the moment (e.g. proceed with touching your face, or stop face-touching and take an alternative behavior).
  Arms: Mindfulness-based "STOP touching your face" intervention

SUMMARY:
This single-blind, randomized, controlled, trial is to assess the efficasy of a brief mindfulness-based "STOP touching your face" training program to reduce or avoid face-touching to low people's chances of catching infectious diseases like COVID-19.

DETAILED DESCRIPTION:
Background Face-touching behavior often happens frequently and automatically, and poses potential risk for spreading infectious disease. Mindfulness-based interventions (MBIs) have shown its efficacy in the treatment of behavior disorders. This study aims to evaluate an online mindfulness-based brief intervention skill named "STOP (Stop, Take a Breath, Observe, Proceed) touching your face" in reducing face-touching behavior.

Methods This will be a single-blind, randomized, controlled, trial. We will recruit 1,000 participants, and will randomize and allocate participants 1:1 to the "STOP touching your face" intervention group (n=500) and the control group (n=500). All participants will be asked to monitor and record their face-touching behavior. The intervention group will receive the brief online mindfulness-based "STOP touching your face" program, and the control group will receive control intervention. Primary outcome will be the efficacy of short-term mindfulness-based "STOP touching your face" intervention for reducing the frequency of face-touching. The secondary outcomes will be the reduction of the duration of face-touching after intervention; the correlation between the psychological traits of mindfulness and face-touching behavior; and the differences of face-touching behavior between left-handers and right-handers. We will recruit 1000 participants from April to June 2020 or until the recruitment process is complete. The follow-up will be completed in June 2020. We expect all trial results to be available by the end of June 2020.

Discussion This is the first RCT to evaluate the efficacy of brief mindfulness intervention to reduce face-touching behavior. We expect that "STOP touching your face" has a significantly greater reduction the frequency of face-touching behavior than the control intervention. As "STOP touching your face" is a brief and simple skill, the public health impact of its expansion world-wide could be enormous, helping us to manage any face-touching spread infectious diseases, like Coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Being able to access online services
3. Being able to read and write in Chinese
4. Expressing an interest in participant this study
5. Willing to provide informed consent to participate in the study

Exclusion Criteria:

1. Under 18 years of age
2. Unable to access online services
3. Unable to read and write in Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Reduction of frequency of face-touching behavior | 2 hours
  This will be calculated as the total times of face-touching (including the eyes, nose, mouth, ears, cheeks, chin, neck, forehead, hair) during a 60-minute period before the intervention minus the total times of face-touching after the intervention.

SECONDARY OUTCOMES:
Reduction of percentage of participants touching their faces | 2 hours
  This will be calculated as the percentage of participants touching their faces (including any of the following areas: the eyes, nose, mouth, ears, cheeks, chin, neck, forehead, hair) during a 60-minute period before the intervention minus the percentage of participants touching their faces after the intervention.
Five Facet Mindfulness Questionnaire (FFMQ) | 2 hours
  To measure the correlation between the psychological traits of mindfulness (measured by FFMQ) and face-touching behavior. The self-report scale of FFMQ is currently the most frequently used mindfulness questionnaire to measure changes in participant's tendency to be mindful in daily life by the following five related facets: observing(noticing, attending to sensations, perceptions, thoughts, feelings; 8 items), describing (labeling feelings, thoughts with words), acting with awareness (automatic pilot, concentration, non-distraction), non-judging internal experience, and non-reactivity to internal experience. Participants will be asked to what extent each of the statements are true of them. Each item is on a 1 to 5 Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true). The factor structure of the short version (FFMQ-15) will be used in this study, which has been consistent with that of the FFMQ-39.
The Edinburgh Handedness Inventory (EHI) | 2 hours
  To measure the differences of face-touching behavior between left-handers and right-handers. EHI is the most widely used 10-item self-report inventory to assess handedness. It is comprised of the following 10 activities: (1) writing, (2) drawing, (3) throwing, (4) using scissors, (5) a toothbrush (6) knife (without fork), (7) spoon, and such activities involving both hands as (8) using a broom (upper hand), (9) striking a match, and (10) unscrewing the lid of a bottle. To complete the EHI, one or two check marks are placed under "left (L)" or "right (R)" columns, indicating strength of preference for each activity. Participants will be asked write "2", "1" or "0" in the appropriate corresponding column. If the preference is very strong that they would never try to use the other hand unless absolutely forced to, then they will mark this column as "2" and the other column as "0". If they are really indifferent, they will mark it as "1" in both columns.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanhui Liao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang J, Wang L, Luo T, Wu S, Wu Z, Chen J, Pan C, Wang Y, Liu Y, Luo Q, Guo X, Xie L, Zhou J, Sun Y, Chen W, Liao Y. Effectiveness of a Brief Mindfulness-Based Intervention of "STOP touching your face" During the COVID-19 Pandemic: a Randomized Controlled Trial. Mindfulness (N Y). 2022;13(12):3123-3133. doi: 10.1007/s12671-022-02019-x. Epub 2022 Nov 9. PMID 36408118
- [Derived] Liao Y, Wang L, Luo T, Wu S, Wu Z, Chen J, Pan C, Wang Y, Liu Y, Luo Q, Guo X, Xie L, Zhou J, Chen W, Tang J. Brief mindfulness-based intervention of 'STOP (Stop, Take a Breath, Observe, Proceed) touching your face': a study protocol of a randomised controlled trial. BMJ Open. 2020 Nov 24;10(11):e041364. doi: 10.1136/bmjopen-2020-041364. PMID 33234653